CLINICAL TRIAL: NCT00129857
Title: Efficacy and Safety Evaluation of a Single Intravenous Dose of Dexanabinol in Patients Suffering From Severe Traumatic Brain Injury
Brief Title: Dexanabinol in Severe Traumatic Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmos (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PH-2000-1
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2004-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — HU 211

INTERVENTIONS:
Drug: Dexanabinol

SUMMARY:
Each year a large number of patients are hospitalized at Shock Trauma Centers with severe head injuries. Bleeding into and swelling of these patients' brains may cause compression of vital structures, disability and death. Sometimes surgery is needed. Unfortunately, the investigators have no medication to treat the bad effects of head trauma. Part of the brain damage is due to toxic chemicals (including one called glutamate) that are released by the damaged nerves. Dexanabinol may prevent some of the bad effects of glutamate on the brain and may protect the brain against uncontrollable swelling and death.

DETAILED DESCRIPTION:
Dexanabinol is a synthetic, non-psychotropic cannabinoid derivative that because of its dextro-configuration is compatible with activation of cannabinoid receptors in the brain. It combines the ability to block NMDA receptors and neuroinflammatory cascades in the same molecule. Dexanabinol scavenges free radicals, protects neurons from toxicity of free radical generators and inhibits lipopolysaccharide-induced production of prostaglandin E2, NO and TNF-a by macrophages in culture.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic head injury within the last 6 hours
* Glasgow Coma Motor score of 2 to 5; severity requires intracranial pressure (ICP) monitoring
* Brain computed tomography (CT) showing intracranial parenchymal abnormality and hemodynamically stable
* An informed consent

Exclusion Criteria:

* Penetrating head injury
* Spinal cord injury
* Coma due to pure epidural hematoma with initial Glasgow Coma Scale (GCS) of => 12
* Previous major cerebral damage
* Concomitant severe conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860
Dates: Start 2001-01; Study Completion 2004-09

PRIMARY OUTCOMES:
Glasgow Outcome Scale Extended (GOSE) at 6 months

SECONDARY OUTCOMES:
GOSE at 3 months
Mortality rates at 10 days and 6 months
Intracerebral pressure during first 72 hours of trauma
Neuroworsening at 10 days
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Maas, M.D., Study Chair — Dept. of Neurosurgery, Dijkzigt Hospital, Rotterdam, Holland

REFERENCES:
- [Result] Maas AI, Murray G, Henney H 3rd, Kassem N, Legrand V, Mangelus M, Muizelaar JP, Stocchetti N, Knoller N; Pharmos TBI investigators. Efficacy and safety of dexanabinol in severe traumatic brain injury: results of a phase III randomised, placebo-controlled, clinical trial. Lancet Neurol. 2006 Jan;5(1):38-45. doi: 10.1016/S1474-4422(05)70253-2. PMID 16361021